CLINICAL TRIAL: NCT01026714
Title: Evaluation of the CYP2C9 Activity With Dried Blood Spots on Filter Paper Obtained With a Simple Finger Prick
Brief Title: CYP2C9 Activity Evaluated With a Simple Finger Prick
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Pr Jules Desmeules, University Hospital, Geneva
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MICRO CYP2C9
Record Dates: First submitted 2009-12-01; First posted 2009-12-04 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Flurbiprofen; Rifampin; Fluconazole

ARMS (3):
- flurbiprofen 50mg po (Experimental)
  Interventions: Drug: flurbiprofen
- flurbiprofen 50 mg po + CYP2C9 inducer (Experimental)
  Interventions: Drug: flurbiprofen, rifampicin
- flurbiprofen 50 mg po + CYP2C9 inhibitor (Experimental)
  Interventions: Drug: flurbiprofen + fluconazole

INTERVENTIONS:
Drug: flurbiprofen — assessment of flurbiprofen plasmatic and capillary rates
  Arms: flurbiprofen 50mg po
Drug: flurbiprofen, rifampicin — assessment of flurbiprofen plasmatic and capillary rates
  Arms: flurbiprofen 50 mg po + CYP2C9 inducer
Drug: flurbiprofen + fluconazole — assessment of flurbiprofen plasmatic and capillary rates
  Arms: flurbiprofen 50 mg po + CYP2C9 inhibitor

SUMMARY:
The cytochrome P450 enzymes (CYP) are the major drug-metabolizing enzyme system in humans. A great inter- individual variability affects the activity of these enzymes, and consequently the plasma drug concentrations resulting in different pharmacodynamic effects and occurrence of effect sides. Environmental factors, diet, drugs or genetics are responsible for this variability. Genetic factors are very important since the majority of these enzymes are highly polymorphic. For example, over 80 CYP2D6 allelic variants have been discovered so far and are associated to the absence, a decrease, or an increase in enzyme activity. Most polymorphisms were detected by adverse reactions occurring in a group within the population after normal doses of drugs had been administrated. Those patients experiencing adverse reactions often had a reduced capability to metabolize certain drugs. In clinical therapy, this variability has important consequences including the lack of response to a treatment and/or adverse drug reactions. In order to reduce these potentially unwanted events possibly leading to sever adverse reactions or death, it might therefore be of decisive interest to be able to assess the activity of these enzymes at the individual level. Two approaches may be used to assess CYPs activities, genotype and phenotype. Genotype is based on DNA analysis and polymorphism detection. Phenotype consists of administration of "model" drug or probe drug metabolized by a specific CYP and a determination of a ratio between the drug and its metabolite in plasma or urine. The principal drawback of the phenotyping methods is the urine collection overnight or at least 8 hours after the administration of probe test. This procedure is very tedious and time consuming for the patient as well as for the medical staff. The test can be performed in plasma or blood 1-2 hours after probe administration. However, this procedure is invasive and needs an important volume of blood (6 ml). Recently, a novel approach has been developed for the quantitative determination of circulating drug concentrations using dried blood spots (DBS) on filter paper obtained with a simple finger prick. Due to the small blood volume required (about 10 µL) compared to conventional sampling, this minimally invasive method provides a patient-friendly alternative for blood collection in patient population where venous sampling is unethical or impossible (pediatrics).

In addition, DBS sampling does not require the use of anticoagulant, plasma separation and decreases contact with infectious material. Furthermore, dried blood spots can be easily stored and shipped to analytical laboratories without using refrigerated devices.

Thanks to the new developments in analytical techniques (mass spectrometry), which permit quantitative analysis from very small volume of blood. DBS sampling represents a powerful tool for the biomedical analyses, particularly in pharmacokinetic studies where several blood samples are needed and for phenotyping procedures.

ELIGIBILITY:
Exclusion Criteria:

* Allergic to the administrated drugs
* Contact lense
* History of peptic ulcer or digestive bleeding
* Long QT
* Impaired hepatic tests (ASAT, ALAT, GGT, BILI)
* Taking drugs interacting with CYP2C9 activity
* Concomitant disease interacting with CYP2C9 activity

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Flurbiprofen plasma and capillary rates in presence/absence of CYP2C9 inhibitor or inducer | 3 singles days spaced out with one week wash-out periods

SECONDARY OUTCOMES:
Correlation between CYP2C9 Genotype and Phenotype | one day

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Geneva, Switzerland